CLINICAL TRIAL: NCT00463073
Title: A Phase II Trial With Cetuximab, Bevacizumab and Irinotecan for Patients With Malignant Glioblastomas and Progression After Radiation Therapy and Temozolamide
Brief Title: Cetuximab, Bevacizumab and Irinotecan for Patients With Malignant Glioblastomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CBI-GBM-01
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Malignant Gliomas
Keywords: Progressive primary Glioblastoma multiforme
MeSH Terms: conditions — Glioma | interventions — Cetuximab; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab
Drug: Bevacizumab
Drug: Irinotecan

SUMMARY:
Irinotecan has demonstrated activity in malignant gliomas in multiple phase II studies. The activity is limited, with an approximately 15 % response rate and a progression-free survival of 3-5 months. Given the synergy between irinotecan and bevacizumab in colorectal cancer, and the high-level expression of vascular endothelial growth factor on malignant gliomas, one would expect synergy between bevacizumab and irinotecan against gliomas. In addition, 40-50 % of GBM have EGFR amplification/mutation making the EGFR an additional target. By combing cetuximab, with irinotecan and bevacizumab, one would expect further response, than irinotecan and bevacizumab alone. In addition, recurrent gliomas have an extremely poor prognosis, so innovative therapies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histological verification of primary GBM
* Recurrence or progression after standard treatment (debulking surgery of possible, radiotherapy and temozolamide within last six months)
* Evidence of measurable recurrent progressive primary GBM (CT/MRI scan)
* PS 0-2 (ECOG scale)
* Age > 18
* Life expectancy > 3 month
* Normal organ function:
* Platelets > 125 x 109/l
* Hemoglobin >6,2 mmol/l
* Leukocytes > 3 x 109/l
* ACN> 1,5 x 109/l
* ASAT and/or ALAT < 3 x upper normal limit
* Bilirubin < 1,5 x upper normal limit
* Creatinine clearance > 45 ml/min
* Creatinine < 1,5 x upper normal limit
* APTT < normal limit
* INR < normal limit
* Cholesterol < 7 mmol/l
* Fertile females must use oral contraceptive, IUD (intrauterine device) or preservatives. Fertile males must use preservatives.

Exclusion criteria:

* Radiotherapy or chemotherapy within the last 4 weeks.
* Co-medication that may interfere with study results; e.g. immunosuppressive agents other than corticosteroids
* Prior EGFR- or VEGFR- based therapy.
* Any condition (medical, social, psychological), which would prevent adequate information and follow-up
* Any other active malignancy or previous malignancies within the last 5 years, except, adequately treated basal or squamous cell carcinoma of the skin, or carcinoma in situ.
* No hypercholesterolemia or hypertriglyceridemia (despite lipid-lowering therapy).
* Any significant cardiac disease (New York Heart Association Class II or greater), arrhythmia, congestive heart failure, acute myocardial infarction within 6 months or unstable angina pectoris.
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis, coagulapathy or taking ASA, NSAIDs or clopidogrel
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0, anticipation of need for major surgical procedure during the curse of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 0
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 month prior to day 0
* History of known HIV, Hepatitis B and Hepatitis C negative
* Any ongoing infection, uncontrolled diabetes mellitus, serious non-healing wound, ulcer or bone fracture
* Pregnancy or breast feeding
* Requires therapeutic anti-coagulation
* Blood pressure > 150/100 mmHG
* Grade 2 or greater proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD., PH.D., Principal Investigator — Rigshospitalet, Dept. of Oncology
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense